CLINICAL TRIAL: NCT07277946
Title: AtraUmatic Laparoscopic HerNia Repair Clinical Investigation to Evaluate the Safety and Performance of The ECLIPSIUM System for Mesh Fixation IDE
Acronym: UNITE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tissium (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PF00006-CLPR-003
Record Dates: First submitted 2025-11-13; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Hernia
Keywords: Ventral Hernia Repair; Hernia; Hernia Repair
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Intervention Model Description: 1:1 randomization, single-blinded
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- ECLIPSIUM System (Experimental): The ECLIPSIUM System is intended for non-penetrating connection and fastening of prosthetic materials, such as composite meshes, to internal soft tissue during minimally invasive hernia repair procedures by coating the prosthetic material with the biodegradable implantable polymer and photoactivating it in situ with a TISSIUM curing light.
  Interventions: Device: ECLIPSIUM® System
- Resorbable tacks (AbsorbaTack/SorbaFix) (Active Comparator): Resorbable tacks are surgical fasteners used to secure a hernia mesh in place. Resorbable tacks are designed to be absorbed by the body over time, gradually losing strength as the tissue ingrowth into the mesh occurs and takes over the support function.
  Interventions: Device: Resorbable tacks (AbsorbaTack/SorbaFix)

INTERVENTIONS:
Device: ECLIPSIUM® System — The ECLIPSIUM® System functions by applying a biodegradable, implantable polymer coating to the prosthetic material under guidance of a template to ensure appropriate application, followed by in situ photo-activation using the TISSIUM curing light to secure the mesh to the abdominal wall.
  Arms: ECLIPSIUM System
Device: Resorbable tacks (AbsorbaTack/SorbaFix) — Resorbable tacks are surgical fasteners used to secure a hernia mesh in place. Resorbable tacks are designed to be absorbed by the body over time, gradually losing strength as the tissue ingrowth into the mesh occurs and takes over the support function.
  Arms: Resorbable tacks (AbsorbaTack/SorbaFix)

SUMMARY:
The primary purpose of this clinical trial is to assess the safety and performance of the ECLIPSIUM device in securing mesh during ventral hernia repair. The study will evaluate whether ECLIPSIUM, a bioresorbable polymer-based fixation device, is effective in reducing the risk of hernia recurrence when compared with bioresorbable tacks. This information will support understanding of ECLIPSIUM's potential clinical benefits in ventral hernia repair.

DETAILED DESCRIPTION:
A prospective, multi-center, randomized, active control, single-blind non- inferiority study designed to evaluate the safety and effectiveness of the ECLIPSIUM® System versus bioresorbable tacks in mesh fixation in patients undergoing laparoscopic intraperitoneal onlay mesh ventral hernia repair procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is 22 years old or older.
2. Patient is willing and able to provide a signed Patient Informed Consent Form.
3. Patient has a single midline primary ventral, umbilical, or incisional hernia;

   a.Hernia Size is 1 -5 cm in diameter (to be confirmed intraoperatively).
4. Patient is scheduled for a laparoscopic IPOM hernia repair.
5. Hernia can be successfully repaired with a single polyester or polypropylene composite mesh with biodegradable coating with at least a 5 cm overlap of the mesh on all sides of the defect (to be confirmed intraoperatively).
6. Female patients must:

   1. Have a negative urine pregnancy test within 3 days before surgery and agree to consistently use an effective method of contraception through completion of study participation.

      OR
   2. Have reached menopause (no menses for 1 year). OR
   3. Have undergone hysterectomy, bilateral oophorectomy, or tubal ligation.
7. Patient is willing and able to follow the study instructions including completion of study procedures, assessments, and visits.

Exclusion Criteria:

1. Patient has a known or suspected hypersensitivity to the constituent polymer of the investigational device, comparator device, mesh, or other surgical products (e.g., sutures).
2. Patient is taking systemic photosensitivity pharmaceutical products at time of informed consent.
3. Patient has a BMI > 40.
4. Patient is a current smoker, defined as self-reporting smoking more than 1 cigarette per day.
5. Patient's hernia is recurrent and/or the patient has a previous midline primary ventral, umbilical, or incisional hernia repair with mesh implantation.
6. Patient has a life expectancy less than 1 year, in the opinion of the Investigator.
7. Patient is unwilling or unable to follow postoperative instructions.
8. Patient is taking systemic immunosuppressive medications, systemic steroids, or chemotherapy at the time of informed consent.
9. Patient is pregnant, plans to become pregnant during the study period, or is breastfeeding.
10. Patient has a diagnosis of Type 1 Diabetes Mellitus.
11. Patient has uncontrolled Type 2 Diabetes Mellitus (HbA1C ≥ 7.0 within 3 months preceding study enrolment).
12. Patient is currently participating in an investigational drug or device study that has not completed the primary outcome or that clinically interferes with this clinical study's outcome (Note: Studies requiring extended follow-up for products that were investigational, but have since become commercially available, are not considered investigational studies).
13. Patient has more than one hernia defect (single hernia defect between 1-5 cm in diameter from outer edged to outer edge to be confirmed intraoperatively).
14. Patient has areas of weakness, independent from the hernia to be treated, in the area covered by mesh or mesh-adjacent tissues (to be confirmed intraoperatively).
15. Patient with a complex hernia, likely not eligible for laparoscopic repair, as determined by the Investigator (ex. small bowel resection; to be confirmed intraoperatively).
16. Patient is scheduled for an additional surgery within 6 weeks after the index-procedure or has undergone surgery within 90 days before the index-procedure.
17. Patient has severe chronic obstructive pulmonary disease.
18. Patient has an ongoing infection (e.g. elevated temperature, elevated white blood count).
19. In the opinion of the Investigator, the patient is not a suitable candidate for the clinical investigation.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Hernia Recurrence at 6 months | 6 months
  Rate of hernia recurrence of the ECLIPSIUM System compared to resorbable tacks at 6 months post-surgery.
Cumulative Incidence of Complications | 12 months
  Safety of the ECLIPSIUM System will be assessed by collecting and analyzing the cumulative incidence of complications (CIC) related to the ECLIPSIUM System including the following complications:
  * Infection
  * Chronic pain (defined as moderate or greater pain lasting more than 3 months) not otherwise specified
  * Impaired/delayed healing at the surgical site (i.e. hernia repair site; example dehiscence)
  * Allergic reaction/hypersensitivity reaction to the constituent polymer of the investigational device
  * Serious Adverse Device Effect (SADEs)

SECONDARY OUTCOMES:
Hernia Recurrence at 12 months | 12 months
  The secondary efficacy outcome of this study is to demonstrate the rate of hernia recurrence of the ECLIPSIUM System is non-inferior compared to resorbable tacks at 12 months post-surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rosen, Principal Investigator — Northwestern University; William Hope, Principal Investigator — New Hanover Regional Medical Center

IPD SHARING:
Plan to Share IPD: No